CLINICAL TRIAL: NCT03081130
Title: Effects of Intravenous Laser Irradiation on Treatment Resistant Thin Endometrium in Women Undergoing Frozen Thawed Embryo Transfer Cycles
Brief Title: Intravenous Laser Irradiation Effect on Treatment Resistant Thin Endometrium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Hsiao-Wen Tsai, Dr. Hsiao-Wen Tsai, Kaohsiung Veterans General Hospital.
Other Study IDs: Laser on thin endometrium
Record Dates: First submitted 2017-03-09; First posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Endometrium; Laser

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intravenous laser irradiation treatment: We will recruit 30 poor ovarian responders and thin endometrium patients and treat with intravenous laser irradiation of blood (ILIB) via an intravenous catheter for irradiation of the blood under a period of 60 minutes for 10 days.
  Interventions: Procedure: Intravenous laser irradiation treatment
- control: We will recruit 30 poor ovarian responders and thin endometrium patients and treat with oral estradiol 8 mg per day and oestrogen gel 4 g per day for 14 days

INTERVENTIONS:
Procedure: Intravenous laser irradiation treatment — control group
  Groups: Intravenous laser irradiation treatment

SUMMARY:
We will recruit 30 poor ovarian responders and thin endometrium patients, aged 35-45 year old, and treat with intravascular laser irradiation of blood (ILIB) via an intravenous catheter for irradiation of the blood under a period of 60 minutes for 10 days. We will evaluate the number and the quality of oocyte retrieved, endometrium thickness and pregnancy rate. The goal of the study is to evaluate whether ILIB is the efficient treatment to improve the ovarian response and the clinical outcome of the poor ovarian responders and thin endometrium patients.

DETAILED DESCRIPTION:
Intravenous laser irradiation of blood (ILIB) is the use of He-Ne laser (632.8 nm) via an intravenous catheter for irradiation of the blood with a lower power of 1-5 milliwatt (mW) and a period of 10-90 minutes to promote functional re-generation mitochondria and pro-oxidant/antioxidant equilibrium in living bodies. ILIB was developed experimentally by the Russian researchers and was introduced into clinical practice in 1981. The treatment with He-Ne laser has been applied on many organs and on the hematologic and immunologic system. Quite a number of both animal and human experiments have demonstrated that ILIB has a wide range of effects, including biostimulation, analgesia, antiallergic effects, immunomodulation, vasodilatation, antihypoxic, anti-oxidant, anti-aging and anti-inflammatory effects. The aid of treatment of acute cerebral infarction, rheumatoid arthritis, arthrosclerosis of the leg, redifferentiation therapy of malignant tumors has been studies for years and over the past 30 years, there are growing studies that has challenging the therapeutic effect of ILIB.

The incidence of poor ovarian responders and thin endometrium patients among infertile women has been estimated at 9-24%. It fact, as a result of a lower number of oocytes retrieved, there are fewer embryos to select and transfer and subsequently these patients have lower pregnancy rates per transfer and lower cumulative pregnancy rates. Despite an enormous number of papers on the topic of poor ovarian response and thin endometrium patients have been published in the literature, so far it has been impossible to identify any efficient treatment to improve the ovarian response and the clinical outcome of this group of patients. In most cases the mechanism involved in follicular depletion is still not clear. Previous studies showed that treatment with anti-oxidants could improve the outcomes of the poor ovarian responders and thin endometrium patients, however, the effect is limited. Since ILIB has anti-aging, anti-oxidant and anti-inflammatory effects, we want to know the effect on the poor ovarian responders and thin endometrium women. Through the lower power of He-Ne laser to promote functional re-generation mitochondria and pro-oxidant/antioxidant equilibrium, poor ovarian responders and thin endometrium women may gain the power to improve the ovarian function and endometrium function and higher the pregnancy rates.

We will recruit 30 poor ovarian responders and thin endometrium patients and treat with intravenous laser irradiation of blood (ILIB) via an intravenous catheter for irradiation of the blood under a period of 60 minutes for 10 days. We will evaluate the number and the quality of oocyte retrieved, endometrium thickness and pregnancy rate. The goal of the study is to evaluate whether ILIB is the efficient treatment to improve the ovarian response and the clinical outcome of the poor ovarian responders and thin endometrium patients.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit 30 poor ovarian responders and thin endometrium patients

Exclusion Criteria:

* women with underlying medical diseases, such as diabetes or hypertension

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We will recruit 30 poor ovarian responders and thin endometrium patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Endometrium thickness | after intervention 1 month and treated with estradiol
  endometrium thickness evaluated by transvaginal sonography after intervention

SECONDARY OUTCOMES:
pregnancy | 4 weeks after embryo transfer
  pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Hao Tsui, Study Director — Department of Obstetrics and Gynecology, Kaohsiung Veterans General Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kudesia R, Kuokkanen S. Thin endometrium after radiation therapy as an unresolved treatment challenge: a case report. Gynecol Endocrinol. 2016 Sep;32(9):701-703. doi: 10.1080/09513590.2016.1177813. Epub 2016 Apr 29. PMID 27129096
- [Background] Lebovitz O, Orvieto R. Treating patients with "thin" endometrium - an ongoing challenge. Gynecol Endocrinol. 2014 Jun;30(6):409-14. doi: 10.3109/09513590.2014.906571. Epub 2014 Apr 2. PMID 24693854
- [Background] Gleicher N, Kim A, Michaeli T, Lee HJ, Shohat-Tal A, Lazzaroni E, Barad DH. A pilot cohort study of granulocyte colony-stimulating factor in the treatment of unresponsive thin endometrium resistant to standard therapies. Hum Reprod. 2013 Jan;28(1):172-7. doi: 10.1093/humrep/des370. Epub 2012 Oct 18. PMID 23081869
- [Background] Kasius A, Smit JG, Torrance HL, Eijkemans MJ, Mol BW, Opmeer BC, Broekmans FJ. Endometrial thickness and pregnancy rates after IVF: a systematic review and meta-analysis. Hum Reprod Update. 2014 Jul-Aug;20(4):530-41. doi: 10.1093/humupd/dmu011. Epub 2014 Mar 23. PMID 24664156
- [Background] Kazemikhoo N, Sarafnejad AF, Ansari F, Mehdipour P. Modifying effect of intravenous laser therapy on the protein expression of arginase and epidermal growth factor receptor in type 2 diabetic patients. Lasers Med Sci. 2016 Nov;31(8):1537-1545. doi: 10.1007/s10103-016-2012-x. Epub 2016 Jul 12. PMID 27406711
- [Background] Momenzadeh S, Akhyani V, Razaghi Z, Ebadifar A, Abbasi M. Evaluation of the Effects of Intravenous and Percutaneous Low Level Laser Therapy in the Management of Shoulder Myofascial Pain Syndrome. J Lasers Med Sci. 2016 Winter;7(1):16-20. doi: 10.15171/jlms.2016.04. Epub 2016 Jan 7. PMID 27330692
- [Background] Rikihisa N, Watanabe S, Satoh K, Saito Y, Sakai H. Photosensitizer Effects of Artificial Red Cells on Dye Laser Irradiation in an Animal Model Assuming Port-Wine Stain Treatment. Plast Reconstr Surg. 2017 Mar;139(3):707e-716e. doi: 10.1097/PRS.0000000000003082. PMID 28234842
- [Background] Dahmardehei M, Kazemikhoo N, Vaghardoost R, Mokmeli S, Momeni M, Nilforoushzadeh MA, Ansari F, Amirkhani A. Effects of low level laser therapy on the prognosis of split-thickness skin graft in type 3 burn of diabetic patients: a case series. Lasers Med Sci. 2016 Apr;31(3):497-502. doi: 10.1007/s10103-016-1896-9. Epub 2016 Feb 11. PMID 26868033